CLINICAL TRIAL: NCT00302393
Title: A PET Study Examining Pharmacokinetics and Dopamine Transporter Receptor Occupancy of Repeat Dosing of OROS® Methylphenidate (CONCERTA®) and Immediate Release Methylphenidate in Healthy Adults
Brief Title: Study Examining Repeat Dosing of OROS® Methylphenidate (CONCERTA®) and Immediate Release Methylphenidate in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Principal Investigator, Thomas J. Spencer, MD, Assistant Director, Pediatric Psychopharmacology Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2005-p-001811
Record Dates: First submitted 2006-03-10; First posted 2006-03-14 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: healthy volunteers
MeSH Terms: interventions — Methylphenidate

ARMS (2):
- IR-MPH (Active Comparator): Immediate Release Methylphenidate administered before PET Scan
  Interventions: Drug: methylphenidate hydrochloride
- Concerta (Active Comparator): OROS Methylphenidate (Concerta) administered before PET Scan
  Interventions: Drug: OROS methylphenidate hydrochloride

INTERVENTIONS:
Drug: OROS methylphenidate hydrochloride — Subjects will be administered a first dose of one of the study treatments at hour 0 and then a second dose of one of the study treatments at hour 4 at each of the four treatment days in a crossover fashion, so that each subject will have received doses of each combination of treatments during the study. Each dose of OROS MPH will be 36 mg which will be supplied as one 36 mg capsules. Study treatments will be administered with water following an overnight fast of at least 8 hours.
  Arms: Concerta
Drug: methylphenidate hydrochloride — Subjects will be administered a first dose of one of the study treatments at hour 0 and then a second dose of one of the study treatments at hour 4 at each of the four treatment days in a crossover fashion, so that each subject will have received doses of each combination of treatments during the study. Each dose of IR MPH will be 20 mg which will be supplied as one 20 mg capsule. Study treatments will be administered with water following an overnight fast of at least 8 hours.
  Arms: IR-MPH

SUMMARY:
There are two specific aims of this study. The first is to document the pharmacokinetics of dopamine transporter (DAT) receptor occupancy of repeated administration of orally administered, therapeutic doses of a short immediate release-methylphenidate hydrochloride (IR-MPH) and a long-acting formulation of MPH (OROS-MPH) using positron emission tomography (PET) scanning with C-11 altropane as the ligand. The investigators hypothesize that central nervous system (CNS) DAT occupancy of the OROS-MPH to IR-MPH sequence will be greater than that of IR-MPH to OROS-MPH sequence at 5 hours after the initial administration and that the CNS DAT occupancy of the other two formulations will be intermediate.

The second aim of this study is to assess whether the abuse liability potential of delayed, repeated administrations of different formulations of MPH is moderated by the oral delivery system in which a delivery system with slower onset may be safer than one with more rapid early release.

DETAILED DESCRIPTION:
ROS-MPH's pharmacokinetic profile uses an increasing delivery of MPH over the day (ascending pharmacokinetic curve). It was designed to replace IR-MPH TID treatment. The main target of MPH in the brain is the dopamine transporter (DAT). We have an exquisitely sensitive methodology to measure DAT occupancy using C-11 Altropane and Positron Emission Tomography (PET). The time course of decay of the C-11 Altropane permits repeated imaging, thus allowing documentation of the pharmacokinetics of DAT receptor occupancy.

We will test all combinations of initial administration and then delayed (repeated) administration of the two formulations: IR-MPH to IR-MPH; IR-MPH to OROS-MPH; OROS-MPH to IR-MPH; and OROS-MPH to OROS-MPH.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent to participate in the study
2. Age: 18 - 55
3. If female, non-pregnant, non-nursing, using an adequate form of birth control or a negative plasma pregnancy test
4. Supine and standing blood pressure within the range 110/60 to 150/90 mmHg
5. Heart rate, after resting for 5 minutes, within the range 46-90 beats/min
6. Subjects who are within 20% of the ideal weight for height
7. Right handed

Exclusion Criteria:

1. Subjects with marked anxiety, tension, and agitation since the drug may aggravate these symptoms
2. Subjects with known hypersensitivity to methylphenidate or other components of Concerta or Ritalin
3. Subjects with glaucoma
4. Subjects with motor tics or with a family history or diagnosis of Tourette's syndrome
5. Subjects treated with monoamine oxidase inhibitors (MAOIs) or within 14 days of discontinuation of treatment with MAOIs
6. Diagnosis of any psychotic disorder, bipolar disorder, severe depression, severe anxiety, or autism. Subjects with mild mood, oppositional, conduct, and anxiety disorders may be permitted to participate if considered appropriate by the investigator.
7. Scores of Baseline Scales:

   * Hamilton Depression Scale > 17 (out of a possible 67 on the 21-item scale) (Hamilton 1960)
   * Beck Depression Inventory > 19 (out of a possible 63 on the 21-item scale) (Beck et al 1961)
   * Hamilton Anxiety Scale > 21 (out of a possible 56 on the 14-item scale) (Hamilton 1959)
8. Diagnosis of ADHD (attention deficit hyperactivity disorder)
9. History of head trauma with loss of consciousness, organic brain disorders, seizures, or neurosurgical intervention
10. Any clinically significant chronic medical condition, in the judgment of the investigator
11. Mental impairment as evidenced by an intelligence quotient (I.Q.) < 75
12. Exposure to dopamine receptor antagonists within the previous three (3) months
13. Exposure to radiopharmaceuticals within four (4) weeks prior to PET scan
14. Subjects receiving psychotropic medication
15. Any clinically significant abnormality in the screening laboratory tests, vital signs, or 12-lead ECG (electrocardiogram), outside of normal limits
16. Any woman of childbearing potential who is seeking to become pregnant or suspects that she may be pregnant
17. Subjects with a known recent history (within the past six [6] months) of illicit drug or alcohol dependence

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-06; Primary Completion 2007-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The DAT receptor occupancy of OROS MPH and MPH IR using PET scanning with C-11 altropane. Objective measures also provided by d and l ritalinic acid and methylphenidate levels at pre-dose, hour 4, 5 and 6. | Eligible subjects will be asked to return to the study center for five study visits.
  The first visit will consist of a baseline PET scan during which no medication will be administered. For the next four study visits, subjects will be administered a first dose of one of the study treatments at hour 0 and then a second dose of one of the study treatments at hour 4. The study visits may be scheduled five to 30 days apart, but each subject must complete the five visits within a ten-week period.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Spencer, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States